CLINICAL TRIAL: NCT05593068
Title: Retrospective Study of Iron Deposits in the Pancreas by MRI Method of Dialysis Patients With Hemosiderosis Iatrogenic
Brief Title: Iron Deposits in the Pancreas by MRI Method of Dialysis Patients With Hemosiderosis Iatrogenic (ERDFP)
Acronym: ERDFP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: ERDFP
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Iron Deposition; Dialysis; Iatrogenic Hemosiderosis
MeSH Terms: conditions — Siderosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dialysed patients with suspicion of hepatic iron: Patients on dialysis at Claude Galien Private Hospital who had one or more MRI scans to monitor possible hepatic iron overload between May 2012 and March 2018.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Pancreatic MRI

SUMMARY:
Recently, a multidisciplinary scientific conference proposed to consider iron overload in dialysis patients as pathological only in the event of demonstration of radiological (in MRI), pancreatic or cardiac ferric deposits.

In this context, the aim of the proposed scientific study is to demonstrate the presence of ferric deposits in the pancreas by T2* MRI in dialysis patients with radiological hepatic iron overload, particularly in cases of moderate and severe iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, over 18 years old
* Patient on hemodialysis or peritoneal dialysis at the Claude Galien Private Hospital
* Patient on dialysis who has undergone one (or more) abdominal MRI for iron quantification
* Patient who has signed a non-objection form for the retrospective use of their MRI, medical and biological data for the purpose of scientific study

Exclusion Criteria:

* Patient who has signed a form to object to the use of their health data
* Pregnant woman
* Poor adherence to the dialytic technique
* Severe cognitive impairment
* Hepatic cirrhosis
* Frank inflammatory syndrome or an active infectious disease
* Genetic hemochromatosis and transfusion hemosiderosis of hemoglobinopathies and hematological diseases
* Recent major bleeding (< 3 months)
* Recent major surgery (< 3 months)
* Transfusion dependence
* Progressive malignant disease
* Pacemakers incompatible with an MRI and metal heart valves

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient on hemodialysis or peritoneal dialysis at Claude Galien Private Hospital. They had to perform an MRI for iron quantification
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Presence of pancreatic iron deposit | 1 day
  Presence of pancreatic iron deposits as a function of hepatic iron level during iron overload in the dialysis patient will be evaluated from the pancreatic iron concentration measured by MRI and expressed by a T2* value in ms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France

REFERENCES:
- [Derived] Rostoker G, Griuncelli M, Francisco S, Loridon C, Languille-Llitjos E, Boulahia G, Cohen Y. Evidence of pancreatic iron deposits and their association with mortality in dialysis-associated iatrogenic hemosiderosis. Clin Kidney J. 2025 Oct 6;18(11):sfaf309. doi: 10.1093/ckj/sfaf309. eCollection 2025 Nov. PMID 41215782